CLINICAL TRIAL: NCT03703973
Title: Correlation Between Postoperative Cognitive Dysfunction and Telomere Length in Patients With Non-cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Han Yuan, Doctor-in-charge of Anesthetist, Xuzhou Medical University
Other Study IDs: POCDLTL
Record Dates: First submitted 2018-09-27; First posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Postoperative Cognitive Dysfunction; Leukocyte Telomere Length
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- study group: 1000 Male and female patients undergoing non-cardiac surgery at the Affiliated Hospital of Xuzhou Medical University [Jiangsu China]. We do the neuropsychological tests, Mini-Mental score examination (MMSE) and olfaction test 1 day before (baseline) and 1 week,3 months,1 year and 3 years after surgery without safety issue.We also measure their preoperative leukocyte telomere length.
  Interventions: Diagnostic Test: Neuropsychology test
- control group: We enroll 50 healthy volunteers and do the neuropsychological tests, Mini-Mental score examination (MMSE) and olfaction test at 1 day (baseline), 1 week, 3 months, 1 year and 3 years without safety issue.
  Interventions: Diagnostic Test: Neuropsychology test

INTERVENTIONS:
Diagnostic Test: Neuropsychology test — We do the neuropsychological tests, Mini-Mental score examination (MMSE) and olfaction test 1 day before (baseline) and 1 week,3 months,1 year and 3 years after surgery without safety issue.

SUMMARY:
To study on the Postoperative Cognitive Dysfunction: Correlations With Leukocyte telomere length。

ELIGIBILITY:
Inclusion Criteria:

* Non-cardiac surgery patients;

  * Age is greater than or equal to 65 years old;

    * Han Nationality, mother tongue is chinese;

      ④The MMSE score:Illiteracy is greater than or equal to 17 points, primary school is greater than or equal to 20 points, higher secondary school is more than 24 points;

      ⑤The Geriatric Depression Scale (GDS) grade 1 or 2;

      ⑥The important function without serious heart, brain, liver, kidney, lung and other organs;
      * The ASA class I or II;

        * The people signed informed consent.

Exclusion Criteria:

* The diagnosis of neurological and psychiatric disorders, such as Alzheimer's disease, Parkinson's syndrome, multiple sclerosis, schizophrenia, depression, etc.; ②Had severe head and face disease, trauma history or history of surgery;

  * Had a history of influenza in 3 weeks; ④The serious body disease and tobacco, wine and other substance abuse history; ⑤The presence of malignant tumor with shorter survival disease.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We included 1000 Male and female patients undergoing non-cardiac surgery and 50 healthy volunteers at the affiliated hospital of Xuzhou Medical University.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
the neuropsychological test to measure cognitive function | 1 day before surgery(baseline)
Mini-Mental score examination [MMSE] used for screening of dementia | 1 day before surgery(baseline)
the leukocyte telomere length | on the surgery day
the neuropsychological test to measure cognitive function | within the first 7 days (plus or minus 2 days) after surgery
Mini-Mental score examination [MMSE] used for screening of dementia | within the first 7 days (plus or minus 2 days) after surgery
the neuropsychological test to measure cognitive function | within the first 3 months (plus or minus 1 month) after surgery
Mini-Mental score examination [MMSE] used for screening of dementia | within the first 3 months (plus or minus 1 month) after surgery
the neuropsychological test to measure cognitive function | within the first 1 year (plus or minus 3 months) after surgery
Mini-Mental score examination [MMSE] used for screening of dementia | within the first 1 year (plus or minus 3 months) after surgery
the neuropsychological test to measure cognitive function | within the first 3 years (plus or minus 1 year) after surgery
Mini-Mental score examination [MMSE] used for screening of dementia | within the first 3 years (plus or minus 1 year) after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia of the Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China